CLINICAL TRIAL: NCT03698513
Title: A Randomized, Cross-over Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986177 (an Oral Antithrombotic) With Single and Dual Antiplatelet Therapy (Aspirin and Clopidogrel) in Healthy Participants
Brief Title: A Study to Assess Administration of an Oral Anti-thrombotic With Antiplatelet Therapy in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV010-034
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — milvexian; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- BMS-986177 + Aspirin + Clopidogrel (Part 1) (Experimental): BMS-986177 200 mg capsule twice daily (days 1-5) + Aspirin 325 mg tablet once daily (days 1-5) + Clopidogrel 300 mg tablet once daily (day 1) then 75 mg tablet once daily (days 2-5)
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin
- BMS-986177 (Part 1) (Experimental): BMS-986177 200 mg capsule twice daily (days 1-5)
  Interventions: Drug: BMS-986177
- BMS-986177 placebo + Aspirin + Clopidogrel (Part 1) (Placebo Comparator): BMS-986177 placebo match capsule twice daily (days 1-5) + Aspirin 325 mg tablet once daily (days 1-5) + Clopidogrel 300 mg once daily (day 1) then 75 mg tablet once daily (days 2-5)
  Interventions: Other: Placebo (for BMS-986177); Drug: Clopidogrel; Drug: Aspirin
- BMS-986177 (Part 2) (Experimental): BMS-986177 200 mg capsule twice daily (days 1-5)
  Interventions: Drug: BMS-986177
- BMS-986177 placebo + Clopidogrel (Part 2) (Placebo Comparator): BMS-986177 placebo match capsule twice daily (days 1-5) + Clopidogrel 300 mg tablet once daily (day 1) then 75 mg tablet once daily (days 2-5)
  Interventions: Other: Placebo (for BMS-986177); Drug: Clopidogrel
- BMS-986177 + Clopidogrel (Part 2) (Experimental): BMS-986177 200 mg capsule twice daily (days 1-5) + Clopidogrel 300 mg tablet once daily (day 1) then 75 mg tablet once daily (days 2-5)
  Interventions: Drug: BMS-986177; Drug: Clopidogrel
- BMS-986177 (Part 3) (Experimental): BMS-986177 200 mg capsule twice daily (days 1-5)
  Interventions: Drug: BMS-986177
- BMS-986177 placebo + Aspirin (Part 3) (Placebo Comparator): BMS-986177 placebo match capsule twice daily (days 1-5) + Aspirin 325 mg tablet once daily (days 1-5)
  Interventions: Other: Placebo (for BMS-986177); Drug: Aspirin
- BMS-986177 + Aspirin (Part 3) (Experimental): BMS-986177 200 mg capsule twice daily (days 1-5) + Aspirin 325 mg tablet once daily (days 1-5)
  Interventions: Drug: BMS-986177; Drug: Aspirin

INTERVENTIONS:
Drug: BMS-986177 — BMS-986177 capsule
  Arms: BMS-986177 (Part 1); BMS-986177 (Part 2); BMS-986177 (Part 3); BMS-986177 + Aspirin (Part 3); BMS-986177 + Aspirin + Clopidogrel (Part 1); BMS-986177 + Clopidogrel (Part 2)
Other: Placebo (for BMS-986177) — BMS-986177 placebo match capsule
  Arms: BMS-986177 placebo + Aspirin (Part 3); BMS-986177 placebo + Aspirin + Clopidogrel (Part 1); BMS-986177 placebo + Clopidogrel (Part 2)
Drug: Clopidogrel — Clopidogrel tablet
  Arms: BMS-986177 + Aspirin + Clopidogrel (Part 1); BMS-986177 + Clopidogrel (Part 2); BMS-986177 placebo + Aspirin + Clopidogrel (Part 1); BMS-986177 placebo + Clopidogrel (Part 2)
Drug: Aspirin — Aspirin tablet
  Arms: BMS-986177 + Aspirin (Part 3); BMS-986177 + Aspirin + Clopidogrel (Part 1); BMS-986177 placebo + Aspirin (Part 3); BMS-986177 placebo + Aspirin + Clopidogrel (Part 1)

SUMMARY:
This study will investigate the safety and interaction of BMS-986177 in healthy volunteers, when administered with Aspirin and/or Clopidogrel

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have a Body Mass Index (BMI) of 18.0 to 32.0 kg/m2, inclusive.
* Must have a normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) of > 80 mL/min/1.73 m2 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula and the absence of protein in the urine

For Parts 1 and 2:

• Must be a clopidogrel responder (eg, a decrease in platelet aggregation of at least 30% after a single 600-mg dose of clopidogrel compared with baseline).

Exclusion Criteria:

* Any significant acute or chronic medical illness, including tinnitus or any other condition listed as a contraindication in the aspirin package insert.
* History of dizziness and/or recurrent headaches (i.e. daily headaches lasting for 1 week's duration in the last month prior to study treatment administration).
* History of head injury in the last 2 years, including participants with base skull fractures, intracranial tumor, or aneurysm.
* History of gastroesophageal reflux disease, dyspepsia (indigestion), protracted nausea, or chronic diarrhea (defined as 3 or 4 loose stools per day that last for ≥ 4 weeks) within the past 6 months.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to Day 33
Incidence of Serious Adverse Events (SAEs) | Up to Day 95
Incidence of Adverse Events (AEs) leading to discontinuation | Up to Day 33
Number of participants with vital sign abnormalities | Up to Day 33
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to Day 33
Number of participants with clinical laboratory abnormalities | Up to Day 33
Number of participants with physical examination abnormalities | Up to Day 33

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 33
  Cmax of BMS-986177, acetylsalicylic acid, salicylic acid, clopidogrel and clopidogrel metabolite
Area under the plasma concentration time curve in one dosing interval [AUC(TAU)] | Up to Day 33
  AUC(TAU) of BMS-986177, acetylsalicylic acid, salicylic acid, clopidogrel and clopidogrel metabolite
Time of maximum observed concentration (Tmax) | Up to Day 33
  Tmax of BMS-986177, acetylsalicylic acid, salicylic acid, clopidogrel and clopidogrel metabolite
Terminal plasma half-life (T-HALF) | Up to Day 33
  T-Half of BMS-986177, acetylsalicylic acid, salicylic acid, clopidogrel and clopidogrel metabolite
Trough observed plasma concentration (Ctrough) | Up to Day 26
  Ctrough of BMS-986177, acetylsalicylic acid, salicylic acid, clopidogrel and clopidogrel metabolite
Apparent total body clearance (CLT/F) | Up to Day 33
  CLT/F of BMS-986177, aspirin, clopidogrel
Volume of distribution (Vz/F) | Up to Day 33
  Vz/F of BMS-986177, aspirin, clopidogrel

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- [Derived] Perera V, Abelian G, Luettgen J, Aronson R, Li D, Wang Z, Zhang L, Lubin S, Merali S, Murthy B. Safety, tolerability, pharmacokinetics and pharmacodynamics of milvexian with aspirin and/or clopidogrel in healthy participants. Sci Rep. 2024 Jul 18;14(1):16591. doi: 10.1038/s41598-024-67182-8. PMID 39025971
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm